CLINICAL TRIAL: NCT00347035
Title: INFLUENCE OF TOPICAL INDOMETHACIN ON HYPOTHENSIVE EFFECT OF BRIMONIDINE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 0771/04
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-10-26 (Estimated); Status verified 2006-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Brimonidine Tartrate

INTERVENTIONS:
Drug: brimonidine

SUMMARY:
Purpose:

To evaluate the influence of the nonsteroidal anti-inflammatory indomethacin on the brimonidine intraocular pressure (IOP) lowering effect.

Methods:

A randomized double-masked study was carried out. Patients medicated with timolol maleate 0,5% and needed complementary medication were random allocated into two groups: (a) brimonidine tartarate 0,15% and indomethacin 1% or (b) brimonidine tartarate and placebo (balanced saline solution). If patient's both eyes were eligible, they were allocated to the same group.

IOP was measured at two weeks, one month and two months after study beginning. The mean IOP of the eyes was used for analyzes, in the case of two eligible eyes. For statistical analyzes repeated measures analysis was used.

ELIGIBILITY:
Inclusion Criteria:

* primary open-angle glaucoma or ocular hypertension patients with the following criteria: 18 years of age or older, insufficient response to monotherapy with timolol maleate 0,5%, and adequate compliance in follow-up treatment

Exclusion Criteria:

* hypersensitivity to eyedrop solutions, insufficient compliance in follow-up treatment, pregnancy or childbearing potential.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Aline K Sousa, MD, Principal Investigator — UNIFESP/EPM Federal University of São Paulo